CLINICAL TRIAL: NCT06152822
Title: Pyrotinib Combined With Capecitabine and Bevacizumab for Patients With HER2 Positive Breast Cancer and Brain Metastases：a Single-arm,Prospective,Phase II Study
Brief Title: Pyrotinib Combined With Capecitabine and Bevacizumab for Patients With HER2 Positive Breast Cancer and Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Tengfei Chao, Tongji Hospital Affiliated of Tongji Medical College Huazhong University of Science and Technology, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20230957
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer With Brain Metastases
Keywords: pyrotinib; capecitabine; bevacizumab; breast cancer; brain metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): pyrotinib+capecitabine+bevacizumab
  Interventions: Drug: pyrotinib+capecitabine+bevacizumab

INTERVENTIONS:
Drug: pyrotinib+capecitabine+bevacizumab — pyrotinib: ≥160mg qd capecitabine: 1000mg/m2,bid,q1-14,q3w bevacizumab:7.5mg/kg,iv,q3w

SUMMARY:
This study intends to conduct a small, prospective, single-center clinical study to explore and evaluate the efficacy and safety of pyrrotinib combined with capecitabine and bevacizumab in HER2-positive advanced breast cancer with brain metastases.The overall objective is to provide a new drug regimen for HER2 positive breast cancer patients with brain metastases by balancing survival benefits and patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. ECOG PS score ≤2
3. Pathologically confirmed advanced breast cancer with positive HER-2 expression;
4. Patients with brain metastases identified by MRI/ enhanced CT with at least one measurable lesion of brain parenchyma according to RECIST 1.1 criteria. There are no requirements as to whether extracranial lesions can be measured.
5. Patients with brain metastases who have not received local treatment in the past and have been treated more than two weeks since the end of the last systemic treatment。Patients with new brain lesions after craniotomy were allowed if they did not receive postoperative radiotherapy and were at least 2 weeks away from surgery.
6. Previous treatment:

   1. Prior treatment with trastuzumab and other HER2-targeting macromolecular antibodies is permitted;
   2. Prior chemotherapy was allowed with any line of chemotherapy. Prior use of endocrine therapy is permitted
   3. Patients who had not previously used capecitabine or progressed after 6 months of discontinuation during metastatic disease or 12 months of discontinuation during adjuvant therapy were admitted.
   4. Concomitant use of bisphosphonates, mannitol, and glucocorticoids was allowed, provided that the glucocorticoid dose was stable for at least a week before enrollment and that the hormone dose was less than 5mg/ day of dexamethasone or equivalent.
7. The expected survival is not less than 6 months.
8. Major organ function is normal, meet the following criteria:

   1. Blood routine: ANC ≥1.0×109/L;PLT ≥100×109/L;Hb ≥90g/L
   2. Blood biochemistry: TBIL ≤1.5 times the upper limit of normal (ULN); ALT and AST≤3 times ULN;For patients with liver metastases, ALT and AST≤5×ULN; BUN and Cr≤1×ULN and creatinine clearance ≥50mL/min (CockcroftGault formula);
   3. Heart color ultrasound: LVEF≥50%;
   4. 12-lead electrocardiogram: Fridericia corrected QT interval (QTcF) < 450ms for males and < 470 ms for females.
9. Voluntarily participate in this study, sign informed consent, have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients with known leptomeningeal metastases, defined as positive imaging or CSF cytology, or clear indications of clinically significant leptomeningeal involvement.
2. need emergency neurosurgery intervention (e.g., removal, shunt placement) of CNS complications.Patients with brain metastases that are poorly controlled by hormonal dehydration and hormonal therapy, such as uncontrollable intracranial hypertension, ejection vomiting, mental disorders, epilepsy, cognitive impairment, etc.
3. There is a third space effusion that cannot be controlled by drainage or other methods (such as excessive pleural fluid and ascites).
4. Patients who had received chemotherapy, surgery or molecular targeted therapy within 2 weeks before enrollment; Patients who received endocrine therapy within 1 week prior to enrollment; Minor procedures such as tumor biopsy, thoracopuncture, or intravenous catheter placement are permitted.
5. Participated in other new drug clinical trials within 4 weeks before enrollment.
6. Have used or currently using tyrosine kinase inhibitors targeting HER-2 (including lapatinib, lenatinib and pyrrotinib, etc.).
7. Other malignancies within the previous 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, or skin squamous cell carcinoma.
8. Receive any other anti-tumor therapy.
9. Have used or currently using bevacizumab
10. There are other concurrent serious and/or uncontrolled conditions that may affect the study, including any of the following:

    1. unable to swallow, chronic diarrhoea and intestinal obstruction, with multiple factors affecting drug use and absorption;
    2. patients with allergy or known history of allergy to the components of this regimen; A history of immunodeficiency, including HIV testing positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
    3. had serious heart disease, including: a.myocardial infarction; b. Heart failure; c.any other heart disease that the investigator determines is not suitable for participation in the study;
    4. infection;
11. Pregnant and lactating women, fertile women who tested positive for baseline pregnancy tests, or women of childbearing age who were unwilling to use effective contraception throughout the trial period.
12. The investigator considers the patient unsuitable for participation in any other circumstances of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate in the CNS | Up to 2 years
  Assess the response rate in the CNS by MRI according to modified Response Assessment in modified RECIST 1.1 criteria. Objective CNS response is defined as at least 30% decrease in the sum of diameters of CNS target lesions in the absence of new lesions (defined as ≥ 6 mm), increased steroid use, progressive neurological symptoms, and progressive extra-CNS disease as assessed by RECIST 1.1. Confirmatory scans are not required.
Time to CNS progression | up to 2 years
  Time to CNS progression will be defined as the time from treatment initiation to documented disease progression (modified RECIST 1.1 criteria) in the CNS

SECONDARY OUTCOMES:
Overall Survival | Up to 3 years
  OS is defined as the time from treatment initiation until death due to any cause
Progression Free Survival | Up to 2 years
  PFS is defined as the time from treatment initiation to documented disease progression
Overall Response Rate | Up to 2 years
  Evaluate systemic ORR defined as partial response or complete response assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Safety | up to 2 years
  Refers to the proportion of patients with a clinically significant adverse event (AE) (ie, leading to treatment modification or discontinuation, patient hospitalization, death, or permanent sequelae) documented in the medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided